CLINICAL TRIAL: NCT04068428
Title: Reproductive Health of Couples of Childbearing Age: a Community Based Prospective Cohort Study
Acronym: ReH-CP
Status: Completed | Type: Observational
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Principal Investigator, Zehong Zhou, Principal Investigator, Guangzhou Women and Children's Medical Center
Other Study IDs: 201925201
Record Dates: First submitted 2019-08-20; First posted 2019-08-28 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Reproductive Health; Time to Pregnancy; Infertility; Risk Factor; Medical Care
Keywords: Reproductive Health; Time to Pregnancy; Infertility; Risk Factor; Assisted Reproductive Technology; Prospective Cohort
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample will be collected from participants who fail to conceive after 12 months of attempts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This community based prospective cohort study was established to investigate the fecundability of couples of childbearing age. Data are collected regarding age, body mass index, education, menstrual regularity as well as childbearing history. Results of routine examination of leucorrhea, blood glucose, liver function of the female spouse, and semen analysis of the male spouse are obtained from the National Free Pre-conception Check-up Projects (NFPCP) in China. Couples recruited will be followed every 6 months for at least 1 year, and their time to pregnancy as well as behavior of seeking medical care would be recorded. Blood sample and/or information of antral follicle count would be collected from participants who fail to conceive after 12 months of attempts.

DETAILED DESCRIPTION:
Infertility is a heavy burden on families, with important implications for individuals and public health. In the last decades, the trend of delaying marriage and childbearing has further exacerbated the burden of infertility. From February 2010 to November 2011, a large-scale population-based cross-sectional study was conducted in northern and eastern China. It was reported that the overall prevalence of infertility was 15.5% among women 'at risk' of pregnancy, and 25.0% among women attempting to become pregnant in China. The prevalence of infertility was surprisingly high and aroused our great attention. To further explore the fecundability and associated risk factors in current China, this community based prospective cohort study was established. Recruitment will be performed at cites of National Free Pre-conception Check-up Projects (NFPCP). Besides of the information of sociodemographic characteristics and childbearing history of couples, their results of check-ups will also be obtained. By regular follow-ups, valid data of time to pregnancy will be collected. A prospective cohort would provide an opportunity to reveal the incidence of infertility, and explore the underlying risk factors of infertility, as well as the demand of assisted reproductive technology.

ELIGIBILITY:
Inclusion Criteria:

* Couples who finish the national free pre-conception check-up
* Couples who agree to receive follow-ups every half year for at least 1 year

Exclusion Criteria:

* None

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Couples of childbearing age from the cites of National Free Pre-conception Check-up Projects (NFPCP) in city of Guangzhou in Guangdong Province, or the city of Haikou in Hainan Province, will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 2313 (Actual)
Dates: Start 2019-07-26 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Time to pregnancy | From date of recruitment until the date of last menstrual period when conceived, assessed up to 1 year
  Assessed by calculate the intervals between last menstrual period when conceived and the timing of termination of contraception.

SECONDARY OUTCOMES:
Prevalence of infertility | After 1 year of follow-up
  Infertility was defined according to the World Health Organization manual as failing to achieve pregnancy after at least 12 months of unprotected regular sexual intercourse.

CONTACTS AND LOCATIONS:
Overall Officials: Zehong Zhou, MD, Principal Investigator — Guangzhou Women and Children's Medical Center, China
Locations (4):
- China (4):
  - Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong
  - Tianhe District Maternal and Child Health Hospital, Guangzhou, Guangdong
  - Longhua District Maternal and Child Health Hospital, Haikou, Hainan
  - Qiongshan District Maternal and Child Health Hospital, Haikou, Hainan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou Z, Zheng D, Wu H, Li R, Xu S, Kang Y, Cao Y, Chen X, Zhu Y, Xu S, Chen ZJ, Mol BW, Qiao J. Epidemiology of infertility in China: a population-based study. BJOG. 2018 Mar;125(4):432-441. doi: 10.1111/1471-0528.14966. Epub 2017 Dec 28. PMID 29030908